CLINICAL TRIAL: NCT04647019
Title: The Effects of Wild Blueberries on Depressive Symptoms in Young Adults: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: The Effects of Wild Blueberries on Depressive Symptoms in Young Adults
Acronym: BluMood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Wild Blueberry Association of North America (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20/13
Record Dates: First submitted 2020-10-21; First posted 2020-11-30 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Depression; Anxiety; Anhedonia
Keywords: Blueberry; Anthocyanins
MeSH Terms: conditions — Depression; Anxiety Disorders; Anhedonia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry powder (Experimental)
  Interventions: Dietary Supplement: Wild blueberry powder
- Placebo powder (Experimental)
  Interventions: Dietary Supplement: Placebo powder

INTERVENTIONS:
Dietary Supplement: Wild blueberry powder — 22 g freeze-dried wild blueberry (Vaccinium angustifolium) powder consumed daily with 250 ml water. The powder is sealed in sachets and stored at -24 °C, except when transported. Participants are asked to store the sachets in a freezer until consumption.
  Arms: Blueberry powder
Dietary Supplement: Placebo powder — 22 g placebo powder matched for macronutrients, color, and flavor consumed daily with 250 ml water. The powder is sealed in sachets and participants are asked to store the sachets in a freezer until consumption.
  Arms: Placebo powder

SUMMARY:
This study aims to investigate the effects of a 6-week dietary intervention of 22 g freeze-dried whole wild blueberry powder. The outcomes include measures of depression, anxiety, anhedonia, cognitive function, and biomarkers of inflammation and oxidative stress.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, parallel-design study assessing the effects of a 6-week intervention of wild blueberry powder in young adults with depressive symptoms. A total of 60 participants will be randomly assigned to either 22 g blueberry powder or a matched placebo powder consumed daily with water. The severity of depression, anxiety, anhedonia, perceived stress, and quality of life will be measured at baseline and 6 weeks later. In addition, we will assess changes in cognitive function and transient mood 2 hours after consuming a single dose of blueberries.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 24 years of age
* Patient Health Questionnaire-9 score ≥ 10 and a score ≥ 2 on the sum of items 1 and 2
* Willingness to provide blood samples

Exclusion Criteria:

* Any medically significant condition (e.g. diabetes, endocrine or gastrointestinal disorders)
* Taking medication (excluding hormonal contraception)
* History of mental illness (excluding anxiety and unipolar depressive disorders)
* Allergy to blueberries or any other Vaccinium species
* Receiving psychotherapy or counselling

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | 6 weeks
  A validated 21-item self-rated scale for assessing depression severity. The scale ranges from 0 to 63 points with higher scores indicating more severe depressive symptomatology.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 6 weeks
  A self-rated scale of depressive symptoms. The scale ranges from 0 to 27 points with higher scores indicating more severe depression.
Generalized Anxiety Disorder 7-item Scale (GAD-7) | 6 weeks
  A brief self-rated scale of generalized anxiety. The scale ranges from 0 to 21 points with higher scores indicating more severe anxiety.
Snaith-Hamilton Pleasure Scale (SHAPS) - modified version | 6 weeks
  A 14-item self-rated scale for measuring anhedonia. Each item has been modified to have five possible responses, which are scored as follows: "strongly disagree" (4 points), "somewhat disagree" (3 points), "neither agree nor disagree" (2 points), "somewhat agree" (1 point), "strongly agree" (0 points). Thus, the scale will range from 0 to 56 points with higher scores indicating greater levels of anhedonia.
Perceived Stress Scale (PSS-10) | 6 weeks
  A validated 10-item questionnaire to measure levels of perceived stress. The scale ranges from 0 to 40 points with higher scores indicating greater stress levels.
Composite Quality of Life Index | 6 weeks
  A 44-item composite index of quality of life derived by adding 11 facets of the WHOQOL-100 Questionnaire (General Health and Life Satisfaction, Pain and Discomfort, Energy and Fatigue, Sleep and Rest, Positive Feelings, Cognitive Function, Self-esteem, Negative Feelings, Activities of Daily Living, Work Capacity, and Personal Relationships). The scale ranges from 0 to 176 points with higher scores indicating better quality of life.
Positive affect as measured by PANAS-X | 2 hours post-ingestion
  Positive affect will be calculated by adding the values of the 21 positive items of the Positive and Negative Affect Schedule-X and the additional item "motivated". Thus, the scale will range from 0 to 88 points with higher scores indicating better mood.
Positive affect as measured by PANAS-X | 6 weeks
  Positive affect will be calculated by adding the values of the 21 positive items of the Positive and Negative Affect Schedule-X and the additional item "motivated". Thus, the scale will range from 0 to 88 points with higher scores indicating better mood.
Negative affect as measured by PANAS-X | 2 hours post-ingestion
  Negative affect will be calculated by adding the values of the 25 negative items of the Positive and Negative Affect Schedule-X. Thus, the scale will range from 0 to 100 points with higher scores indicating worse mood.
Negative affect as measured by PANAS-X | 6 weeks
  Negative affect will be calculated by adding the values of the 25 negative items of the Positive and Negative Affect Schedule-X. Thus, the scale will range from 0 to 100 points with higher scores indicating worse mood.
Cognitive flexibility | 2 hours post-ingestion
  A task-switching test will be used to assess cognitive flexibility when switching between two predictable tasks requiring simple numerical decisions. The main outcome of interest is the average accuracy (0 to 100%).
Cognitive flexibility | 6 weeks
  A task-switching test will be used to assess cognitive flexibility when switching between two predictable tasks requiring simple numerical decisions. The main outcome of interest is the average accuracy (0 to 100%).
Brain-derived neutrophic factor (BDNF) in serum | 6 weeks
  Serum levels of BDNF will be analyzed using enzyme-linked immunosorbent assay (ELISA).
Interleukin-6 (IL-6) in serum | 6 weeks
  Serum levels of IL-6 will be analyzed using enzyme-linked immunosorbent assay (ELISA) as a marker of systemic inflammation.
C-reactive protein (CRP) in serum | 6 weeks
  Serum levels of CRP will be measured using an automated chemistry analyzer as a marker of systemic inflammation.
Uric acid in serum | 6 weeks
  Serum levels of uric acid will be measured using an automated chemistry analyzer.
Serum total antioxidant capacity (TAC) | 6 weeks
  The total antioxidant capacity (TAC) of serum will be measured to assess systemic antioxidant status.
Serum superoxide dismutase (SOD) | 6 weeks
  Serum levels of superoxide dismutase (SOD) will be measured as an indicator of oxidative stress.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Williams, Professor, Principal Investigator — University of Reading
Locations (1):
- School of Psychology and Clinical Languages, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be made available on a platform such as Open Science Framework (www.osf.io) or a data repository linked to academic journals, in accordance with Open Science principles.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Velichkov M, Bezur Z, van Reekum CM, Williams CM. A biphasic response to blueberry supplementation on depressive symptoms in emerging adults: a double-blind randomized controlled trial. Eur J Nutr. 2024 Jun;63(4):1071-1088. doi: 10.1007/s00394-023-03311-9. Epub 2024 Feb 1. PMID 38300292

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT04647019/Prot_SAP_001.pdf